CLINICAL TRIAL: NCT05527561
Title: Effect of Latin Dance on Social Physique Anxiety and Physical Self-esteem of Middle School Girls
Brief Title: Effect of Latin Dance on Middle School Girls' Social Physique Anxiety and Physical Self-esteem
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Liu Xutao, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: Liu Xutao
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Mental Health Issue; Physical Illness
Keywords: Latin dance; Social physique anxiety; Physical self-esteem

STUDY DESIGN:
Intervention Model Description: In this experiment, the experimental group conducted the Latin dance training content intervention designed in this study. In contrast, the control group will exercise basketball training content intended.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Latin Dance-Rumba (Experimental): Rumba dance training was shown for the 1-6 weeks.
  Interventions: Behavioral: Latin dance: Rumba; Behavioral: Latin dance: Cha Cha Cha
- Latin Dance-Cha Cha Cha (Experimental): Cha Cha Cha dance training for the 7-12 weeks.
  Interventions: Behavioral: Latin dance: Rumba; Behavioral: Latin dance: Cha Cha Cha

INTERVENTIONS:
Behavioral: Latin dance: Rumba — Latin dance is a kind of sports dance, which originated in Latin America, includes the rumba, samba, Cha Cha Cha, bullfighting dances and cowboy dances. The intensity of the training is increasing in the first 20 minutes, and the intensity is gradually decreasing in the next 5 minutes.
Behavioral: Latin dance: Cha Cha Cha — Latin dance is a kind of sports dance, which originated in Latin America, includes the rumba, samba, Cha Cha Cha, bullfighting dances and cowboy dances. The intensity of the training is increasing in the first 20 minutes, and the intensity is gradually decreasing in the next 5 minutes.

SUMMARY:
Latin dance is a kind of sports dance, which originated in Latin America, includes the rumba, samba, Cha Cha Cha, bullfighting dances and cowboy dances. Latin dance has bright and strong music rhythm, passion, bold, romantic style, Latin dance has a positive effect on physical and mental health. Latin dance offers a unique dimension that traditional aerobic exercise does not, namely interpersonal communication and interactivity. Dancing may provide additional cognitive benefits compared to other forms of PA, such as walking. Latin dance also provides a unique dimension that traditional aerobic exercise does not, that is, it is a complex sensory-motor rhythmic activity that integrates a variety of physical, cognitive and social factors. Based on the unique charm of Latin dance and previous articles on the influence of dance on social physique anxiety and physical self-esteem, there are few articles on Latin dance, and none of them have studied the influence of Latin dance on these two variables. This study analyzes the Latin dance on the social physique anxiety and physical self-esteem of middle school girls and provides theoretical support for the study to improve the social physique anxiety and physical self-esteem of middle school students, as well as to promote Latin dance. To promote the diversification of Chinese middle school sports in dance teaching.

DETAILED DESCRIPTION:
In the study, the experimental group conducted the 12-week Latin dance training content intervention designed in this study. In contrast, the control group discussed with the teacher and studied the 12-week basketball training content intended. Students participated in a dance exercise program consisting of 40min twice a week (Totally 80 minutes). Control and experimental groups answered SPAS and PSPP questionnaires in the first week. After a 12-week dance training program, both groups were asked to answer SPAS and PSPP questionnaires. Rumba dance training was shown for the first six weeks; Cha Cha Cha dance training for the last six weeks.

Content of Experimental Group:

Week 1: Introduces the classification of Latin dance, starting from the cha-cha dance, telling its origin, music rhythm and dance style characteristics; Week 2: Practice basic standing posture, cha-cha basic frame and hand exercises; Week 3: Reviewed the basic frame and hand shape, introduced the basic step, cha-cha forward and backward step, time step, square step; Week 4: Learn the New York step and the combination of the basic steps of the cha-cha; Week 5: Learn the cha-cha step and the cha-cha turn; Week 6: Learn the basic set combinations of cha-cha; Week 7: Review all the learning material and introduce rumba; Week 8: Learning the basic hand and foot shapes of rumba dance; Week 9: Learning "8" twist hips; Rumba in place change of weight and time step; Week 10: Review the place change of weight and time step, learn rumba forward and backward step, square step; Week 11: Review forward and backward steps, learn rumba New York step and hand step; Week 12: Learning rumba basic set combinations.

ELIGIBILITY:
Inclusion Criteria:

* The population must be middle school girls and between the ages of 13 and 15;
* Contestants must be in good health, but must not have a Latin dance background;
* Only students who can complete these training requirements can be included in the research data.

Exclusion Criteria:

* Boys in middle school should be excluded from this study;
* Some girls' students with professional dance foundation should be excluded;
* Participants were not healthy middle school students such as patients, mental patient, drug addiction, or special students who were seriously depressed, sub-health;
* Students who are consistently late or absent from training sessions will eventually be excluded.

Ages: 13 Years to 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-12-25 (Estimated); Study Completion 2023-01-20 (Estimated)

PRIMARY OUTCOMES:
Social physique anxiety performance of middle school girls | Pretest: Before experiment
  Test by Social Physique Anxiety Scale (SPAS). The Social Physique Anxiety Scale (SPAS) was employed to measure Social physique anxiety. The respondents are asked to rate 12 statements on a 5-point Likert type scale. The anchors are 'not at all' (1), 'slightly' (2), 'moderately' (3), 'very' (4), and 'extremely' (5). Examples of items are: 'I am comfortable with the appearance of my physique' and 'Unattractive features of my physique/figure make me nervous in certain social settings'. Previous research with SPAS has demonstrated test-retest reliability and internal consistency with Cronbach's alpha values of around 0.90.
Physical self-esteem performance of middle school girls | Pretest: Before experiment
  Test by Physical Self-perception Profile (PSPP). The Physical Self-perception Profile (PSPP) is a 30-item self-report questionnaire consisting of five sub-domains, each of which has six items. The sub-domains are: Perceived (1) Sport Competence (Sport), (2) Physical Conditioning (Condition), (3) Bodily Attractiveness (Body), (4) Physical Strength (Strength), and (5) Physical Self-Worth (PSW). Two alternative statements or descriptions of people are presented, from which the individuals can choose the one which best describes themselves, ranging from 'sort of true' to 'really true'. Each item is then scored from 1 to 4.

SECONDARY OUTCOMES:
Social physique anxiety performance of middle school girls | Mid-test: 6 weeks end
  Test by Social Physique Anxiety Scale (SPAS). The Social Physique Anxiety Scale (SPAS) was employed to measure Social physique anxiety. The respondents are asked to rate 12 statements on a 5-point Likert type scale. The anchors are 'not at all' (1), 'slightly' (2), 'moderately' (3), 'very' (4), and 'extremely' (5). Examples of items are: 'I am comfortable with the appearance of my physique' and 'Unattractive features of my physique/figure make me nervous in certain social settings'. Previous research with SPAS has demonstrated test-retest reliability and internal consistency with Cronbach's alpha values of around 0.90.
Physical self-esteem performance of middle school girls | Mid-test: 6 weeks end
  Test by Physical Self-perception Profile (PSPP). The Physical Self-perception Profile (PSPP) is a 30-item self-report questionnaire consisting of five sub-domains, each of which has six items. The sub-domains are: Perceived (1) Sport Competence (Sport), (2) Physical Conditioning (Condition), (3) Bodily Attractiveness (Body), (4) Physical Strength (Strength), and (5) Physical Self-Worth (PSW). Two alternative statements or descriptions of people are presented, from which the individuals can choose the one which best describes themselves, ranging from 'sort of true' to 'really true'. Each item is then scored from 1 to 4.

OTHER OUTCOMES:
Social physique anxiety performance of middle school girls | Post-test: 12 weeks end
  Test by Social Physique Anxiety Scale (SPAS). The Social Physique Anxiety Scale (SPAS) was employed to measure Social physique anxiety. The respondents are asked to rate 12 statements on a 5-point Likert type scale. The anchors are 'not at all' (1), 'slightly' (2), 'moderately' (3), 'very' (4), and 'extremely' (5). Examples of items are: 'I am comfortable with the appearance of my physique' and 'Unattractive features of my physique/figure make me nervous in certain social settings'. Previous research with SPAS has demonstrated test-retest reliability and internal consistency with Cronbach's alpha values of around 0.90.
Physical self-esteem performance of middle school girls | Post-test: 12 weeks end
  Test by Physical Self-perception Profile (PSPP). The Physical Self-perception Profile (PSPP) is a 30-item self-report questionnaire consisting of five sub-domains, each of which has six items. The sub-domains are: Perceived (1) Sport Competence (Sport), (2) Physical Conditioning (Condition), (3) Bodily Attractiveness (Body), (4) Physical Strength (Strength), and (5) Physical Self-Worth (PSW). Two alternative statements or descriptions of people are presented, from which the individuals can choose the one which best describes themselves, ranging from 'sort of true' to 'really true'. Each item is then scored from 1 to 4.

CONTACTS AND LOCATIONS:
Overall Officials: Xutao Liu, PhD, Principal Investigator — University Putra Malaysia
Locations (1):
- Shanghai United International School, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Since this is my doctoral thesis experiment, I won't share it until I graduate.

REFERENCES:
- [Background] Kandola A, Ashdown-Franks G, Hendrikse J, Sabiston CM, Stubbs B. Physical activity and depression: Towards understanding the antidepressant mechanisms of physical activity. Neurosci Biobehav Rev. 2019 Dec;107:525-539. doi: 10.1016/j.neubiorev.2019.09.040. Epub 2019 Oct 2. PMID 31586447
- [Background] Aguinaga S, Marquez DX. Impact of Latin Dance on Physical Activity, Cardiorespiratory Fitness, and Sedentary Behavior Among Latinos Attending an Adult Day Center. J Aging Health. 2019 Mar;31(3):397-414. doi: 10.1177/0898264317733206. Epub 2017 Sep 27. PMID 29254398
- [Background] Hagger MS, Stevenson A. Social physique anxiety and physical self-esteem: gender and age effects. Psychol Health. 2010 Jan;25(1):89-110. doi: 10.1080/08870440903160990. PMID 20391209
- See also: This article is from National Library of Medicine. — https://pubmed.ncbi.nlm.nih.gov/31586447/
- See also: This article is from National Library of Medicine. — https://pubmed.ncbi.nlm.nih.gov/29254398/
- See also: This article is from National Library of Medicine. — https://pubmed.ncbi.nlm.nih.gov/20391209/